CLINICAL TRIAL: NCT06890013
Title: Identifying the Role of Flow Mediated Dilatation Assessment in Acute Coronary Syndromes - Evaluation of the Cor-IS Technology (the FLARE-ACS Trial)
Brief Title: A Prospective, Single-center, Observational Study Aiming to Assess the Predictive Role of Flow Mediated Dilatation in Acute Coronary Syndromes, Combined With Echocardiographic and Biochemical Indices: The Novel Cor-IS Technology Will Also be Evaluated
Acronym: FLARE-ACS
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: 198/31.5.2024
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Acute Coronary Syndromes; Flow Mediated Dilation; Endothelial Function (FMD)
Keywords: acute coronary syndrome; endothelial dysfunction; biomarker; flow mediated dilatation
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 40 ml plasma specimen (-80 grades Celsius)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: Patients hospitalized due to acute coronary syndromes (STEMI, NSTEMI)
  Interventions: Diagnostic Test: Observation group

INTERVENTIONS:
Diagnostic Test: Observation group — Patients with acute coronary syndrome undergo endothelial function assessment using two methods (flow mediated dilatation of the brachial artery and Cor-Is technology) transthoracic echocardiogram and plasma biomarkers' measurement.

SUMMARY:
A prospective, single-center, observational study aiming to assess the predictive role of flow mediated dilatation in acute coronary syndromes, combined with echocardiographic and biochemical indices. The novel Cor-IS technology will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients hospitalized due to acute coronary syndrome (STEMI, NSTEMI)
3. Capability of providing written informed consent
4. Patients able to comply with the follow-up schedule of the study

Exclusion Criteria:

1. Patients with acute coronary syndromes classified as MINOCA, or type II myocardial infarction
2. Patients with rare acute coronary syndrome types, such as spontaneous coronary artery dissection or Takotsubo syndrome
3. Patients with congenital heart disease
4. Age > 85 years
5. Patients with end stage chronic kidney disease
6. Patients with active malignancy or autoimmune diseases which limit their survival
7. Patients with expected survival < 1 year due to other reasons
8. Suboptimal echocardiographic windows
9. Inability to provide written consent
10. Inability to comply with the follow-up schedule of the study
11. Pregnancy
12. Use of intravenous drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized due to acute coronary syndromes (STEMI, NSTEMI) are considered eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Brachial artery endothelial function assessment using the Cor-IS method compared to FMD | 12 months
  The primary outcome of the study is the assessment of brachial artery endothelial function in the therapeutic approach using the Cor-IS method compared to the reference method FMD. The indices of the FMD method (FMD%, shear rate, and FMD/shear) will be compared with the R index of the Cor-IS method at the study's baseline and during follow-up.

SECONDARY OUTCOMES:
FMD% index and MACE | 12 months
  Correlation of the FMD% index with the 3-point MACE (cardiovascular death, non-fatal acute myocardial infarction, stroke)
R-index and MACE | 12 months
  Correlation of the R-index with the 3-point MACE (cardiovascular death, non-fatal acute myocardial infarction, stroke).
FMD% index and rehospitalizations for angina | 12 months
  Correlation of the FMD% index with the total rehospitalizations for angina.
R-index and rehospitalizations for angina | 12 months
  Correlation of the R-index with the total rehospitalizations for angina.
FMD% index and need for revascularization | 12 months
  Correlation of the FMD% index and need for revascularization within 1 year from study enrollment.
R-index and need for revascularization | 12 months
  Correlation of the R-index and need for revascularization within 1 year from study enrollment.
FMD% index and heart failure | 12 months
  Correlation of the FMD% index and the development of heart failure within 1 year from study enrollment.
R-index and heart failure | 12 months
  Correlation of the R-index and the development of heart failure within 1 year from study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Christodoulos E. Papadopoulos, PhD, Principal Investigator — Aristotle University of Thessaloniki, Greece; Georgios Zormpas, MD, Principal Investigator — Aristotle University of Thessaloniki, Greece
Locations (1):
- Ippokratio General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided